CLINICAL TRIAL: NCT04007237
Title: The Comparative Assessment of Mycological Efficacy, Safety, Recurrence, and Cost-effectiveness of Selenium Sulfide 1.8% Shampoo Versus Ketoconazole 2% Shampoo in Pityriasis Versicolor: a Double-blind Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fariz Nurwidya, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: efficacy - PV
Record Dates: First submitted 2019-06-15; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Pityriasis Versicolor
Keywords: mycological efficacy; ketoconazole; selenium disulfide 1,8%; Pityriasis versicolor
MeSH Terms: conditions — Tinea Versicolor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind randomized clinical trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Selsun Shampoo (SeS2 shampoo) (Experimental): Subject were given the SeS2 1.8% shampoo for 2 weeks. They should use it everyday, 10ml each time for 10 minutes. Evaluation was weekly and note for side effects and compliance
  Interventions: Drug: shampoo with different composition
- Ketoconazole shampoo (Active Comparator): Subject were given the Ketoconazole 2% shampoo for 2 weeks. They should use it everyday, 10ml each time for 10 minutes. Evaluation was weekly and note for side effects and compliance
  Interventions: Drug: shampoo with different composition

INTERVENTIONS:
Drug: shampoo with different composition — To reveal the mycological efficacy, safety, recurrence and cost-effectiveness of selenium sulfide 1.8% shampoo (SeS2) and ketoconazole 2% shampoo in the treatment of pityriasis versicolor.

SUMMARY:
There are several topical treatment for Pityriasis Versicolor including ketoconazole and selenium sulfide. Ketoconazole is a broad spectrum anti-fungal drug from imidazole group that has been reported to be effective in PV. The study aimed to reveal the mycological efficacy, safety, recurrence and cost-effectiveness of selenium sulfide 1.8% shampoo (SeS2) and ketoconazole 2% shampoo in the treatment of pityriasis versicolor. A double blind randomized controlled trial was performed in patients with PV during September-December 2018. Patients who involved in this study were allocated to SeS2 or ketoconazole 2% based on block randomization. Physical examinations, scale provocation test, Wood lamp and potassium hydroxide (KOH) examination were conducted to evaluate the treatment response and side effects on 7th - 14th day. Intention to treat analysis was performed in this study. cost-effectiveness was analyzed by Incremental Cost-Effectiveness Ratio (ICER).

ELIGIBILITY:
Inclusion Criteria:

* Having PV characteristic skin lesions,proven by 20% KOH scraping test and Parker Blue-Black® ink, with the founding of short hyphae and group spores or short hyphae only
* willing to participate in the study by signing the written informed consent
* Subjects under the age of 18 with permission from parents or guardians.

Exclusion Criteria:

* A history of hypersensitivity to the ingredients of the shampoo tested.
* Having skin abnormalities with impaired skin integrity
* In the treatment of topical anti-fungal therapy for less than two weeks or systemic anti-fungal for less than one month.
* Pregnancy and breastfeeding.
* Patients with PV lesions on the face.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
mycology efficacy | 7 days
  skin scrapping with KOH test 20% and Parker Blue-Black® ink with the founding of short hyphae and group spores or short hypha only as a positive result
mycology efficacy | 14 days
  skin scrapping with KOH test 20% and Parker Blue-Black® ink with the founding of short hyphae and group spores or short hypha only as a positive result
compliance | 7 days
  the number of day in which a participant using the shampoo which was assigned for minimum 5 days or more and the remaining volume of shampoo does not exceed 25 ml.
compliance | 14 days
  the number of day in which a participant using the shampoo which was assigned for minimum 5 days or more and the remaining volume of shampoo does not exceed 25 ml.
side effect | 7 days
  based on clinical symptoms : itching, burning or stinging sensation. Assessed based on patient records in the diary and through interviews during control
side effect | 14 days
  based on clinical symptoms : itching, burning or stinging sensation. Assessed based on patient records in the diary and through interviews during control
cost-effectiveness | two weeks
  Cost calculations include administrative fees (registration and consultation of doctors), laboratory examinations, medical expenses and compensation for side effects adjusted for the duration of therapy. The results of the calculation of costs obtained are then linked to the negative outcome difference (KOH is still positive) or the value of absolute risk reduction (ARR) on day 14. So that cost efficacy is seen from Incremental Cost-Effectiveness Ratio
recurrence | 1 month
  if the KOH test 20% give a positive result again

CONTACTS AND LOCATIONS:
Locations (1):
- Puskesmas Kecamatan Pulo Gadung, Jakarta, Indonesia